CLINICAL TRIAL: NCT04324268
Title: A Phase 1 Study to Evaluate Safety, Tolerability, and Bioavailability of Subcutaneously Administered Lirentelimab (AK002) in Adult Healthy Volunteers
Brief Title: A Study to Evaluate Safety, Tolerability, and Bioavailability of Subcutaneous Lirentelimab (AK002) in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: AK002-017
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Study Conducted in Healthy Volunteers
MeSH Terms: interventions — AK002

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subcutaneous cohorts will be assigned in a double-blind, randomized, placebo-controlled manner. IV cohorts will be open-label.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- SC 0.3 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive a single dose of 0.3 mg/kg of lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: lirentelimab (AK002)
- SC 1 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive a single dose of 1 mg/kg of lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: lirentelimab (AK002)
- SC 3 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive a single dose of 3 mg/kg of lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: lirentelimab (AK002)
- SC 5 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive a single dose of 5 mg/kg of lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: lirentelimab (AK002)
- IV 1 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive a single dose of 1 mg/kg of lirentelimab (AK002) administered intravenously.
  Interventions: Drug: lirentelimab (AK002)
- IV 3 mg/kg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive a single dose of 3 mg/kg of lirentelimab (AK002) administered intravenously.
  Interventions: Drug: lirentelimab (AK002)
- IV 3 mg/kg of lirentelimab (AK002) (Priming) (Experimental): Subjects in this arm will receive a single dose of 3 mg/kg of lirentelimab (AK002) administered intravenously from an IV bag prepared with extra volume for priming IV set.
  Interventions: Drug: lirentelimab (AK002)
- SC 300 mg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive a single dose of 300 mg of lirentelimab (AK002) administered subcutaneously.
  Interventions: Drug: lirentelimab (AK002)
- SC 450 mg of lirentelimab (AK002) (Experimental): Subjects in this arm will receive a total of 450 mg of lirentelimab (AK002), administered as two separate subcutaneous injections.
  Interventions: Drug: lirentelimab (AK002)

INTERVENTIONS:
Drug: lirentelimab (AK002) — Lirentelimab (AK002) is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8.
  Arms: IV 1 mg/kg of lirentelimab (AK002); IV 3 mg/kg of lirentelimab (AK002); IV 3 mg/kg of lirentelimab (AK002) (Priming); SC 0.3 mg/kg of lirentelimab (AK002); SC 1 mg/kg of lirentelimab (AK002); SC 3 mg/kg of lirentelimab (AK002); SC 300 mg of lirentelimab (AK002); SC 450 mg of lirentelimab (AK002); SC 5 mg/kg of lirentelimab (AK002)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1, single-center study to evaluate safety, tolerability, and bioavailability of subcutaneously administered lirentelimab (AK002) in adult healthy volunteers. Subjects will receive a single dose of intravenous AK002 or subcutaneous lirentelimab (AK002) assigned in a double-blind, randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent.
2. Male or female aged ≥18 and ≤65 years at the time of signing the ICF.
3. Determined by the Investigator to be in good health as documented by medical history, vital signs, physical examination, laboratory assessments, ECG, and by general observations.
4. Subjects must weigh at least 50 kg and have a BMI between 18 g/m2 and 30 kg/m2, inclusive.
5. Negative urine drug screen at Screening.
6. Subjects must have the ability and willingness to attend the necessary visits to the study center and the ability to communicate effectively with the study site personnel.
7. Negative screening ova and parasite test.
8. Female subjects must be either post-menopausal for at least 1 year with FSH level >40 IU/mL at Screening or surgically sterile (tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 3 months, or if of childbearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from Screening until the end of the study, or for 120 days following the last dose of study drug, whichever is longer.
9. Male subjects with female partners of childbearing potential must agree to use a highly effective method of contraception from Screening until the end of the study or for 120 days following the last dose of study drug, whichever is longer. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or late menstrual period) at any time during study participation.

Exclusion Criteria:

1. Peripheral blood absolute eosinophil count >300/µL.
2. Known hypersensitivity to any constituent of the study drug.
3. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study.
4. Presence of abnormal laboratory values considered to be clinically significant by the Investigator.
5. Any disease of condition (medical or surgical) which, in the opinion of the Investigator, would place the subject at increased risk.
6. History of malignancy except carcinoma in situ in the cervix, early stage prostate cancer, or non-melanoma skin cancers.
7. Treatment with chemotherapy or radiotherapy in the preceding 6 months.
8. Treatment for a helminthic parasitic infection within 6 months of screening.
9. Use during the 30 days before Screening (or 5 half-lives, whichever is longer) or use during the Screening period of omalizumab, dupilumab, systemic immunosuppressive drugs, or systemic corticosteroids, except if receiving as part of a premedication protocol.
10. Vaccination with live attenuated vaccines within 30 days prior to initiation of treatment in the study, during the treatment period, or vaccination expected within 5 half-lives (4 months) of study drug administration.
11. Positive hepatitis serology results, except for vaccinated subjects or subjects with past but resolved hepatitis, at Screening.
12. Positive HIV serology results at Screening.
13. Alcohol, drug, or other substance abuse or dependence.
14. Any other reason that, in the opinion of the Investigator or Medical Monitor, makes the subject unsuitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of lirentelimab (AK002) administered subcutaneously by evaluating adverse events assessed using the CTCAE version 5 | Day 0 (baseline) to Day 85
Pharmacokinetics, including bioavailability, of lirentelimab (AK002) administered subcutaneously | Day 0 (baseline) to Day 85

SECONDARY OUTCOMES:
Pharmacodynamics of lirentelimab (AK002) SC formulation as measured by changes in absolute peripheral blood counts of esoinophils | Day 0 (baseline) to Day 85
Bioavailability of lirentelimab (AK002) SC formulation relative to lirentelimab (AK002) IV by analyzing the area under the serum AUC | Day 0 (baseline) to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, PhD, Study Director — Allakos Inc.
Locations (1):
- Allakos Investigational Site, Edgewater, Florida, United States

IPD SHARING:
Plan to Share IPD: No